CLINICAL TRIAL: NCT04748120
Title: Operative vs Non-Operative Management of Acute Appendicitis and Acute Cholecystitis in COVID-19 Positive Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient eligible patients
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Clayton Petro, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-525
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Covid19; Appendicitis; Cholecystitis, Acute; Cholecystitis; Gallstone; Cholecystitis
MeSH Terms: conditions — COVID-19; Appendicitis; Cholecystitis, Acute; Cholecystitis; Gallstones

STUDY DESIGN:
Intervention Model Description: This will be a prospective, non-blinded, pilot randomized controlled trial comparing operative to non-operative management of acute appendicitis and acute cholecystitis in patients with mild to moderate COVID-19 infection. This will be a two-arm trial with intervention 1: intervention 2 allocation ratio of 1:1.
Masking Description: Participants will be informed regarding the treatment they receive at the time of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative management (Active Comparator): Treatment with surgery
  Interventions: Procedure: Operative management
- Non-operative management (Active Comparator): Treatment with antibiotics
  Interventions: Procedure: Non-operative management

INTERVENTIONS:
Procedure: Operative management — Patients will undergo surgical removal of the affected organ. The initial approach will be in a minimally invasive, laparoscopic fashion. If necessary, conversion to an open operation may be performed. These patients will be treated preoperatively and postoperatively with similar antibiotic regimens, however the duration of antibiotic therapies will be dependent on factors such as intraoperative findings, resolution of laboratory abnormalities, and tolerance of oral medications.
  Arms: Operative management
Procedure: Non-operative management — Patients will be treated with 3 days of intravenous antibiotics followed by 7 days of oral antibiotics, as described below:
  Non-penicillin allergic patients
  * piperacillin/tazobactam 3.375g IV every 6 hours for 3 days
  * amoxicillin/clavulanate 875/125mg by mouth every 12 hours for 7 days
  Penicillin allergic patients
  * ertapenem 1g IV every 24 hours for 3 days
  * ciprofloxacin 500mg every 12 hours AND metronidazole 500mg every 8 hours for 7 days
  Patients may be considered to have failed non-operative management (e.g. treatment failure) if they experience absence of clinical improvement, worsening abdominal pain and/or localized/diffuse peritonitis in the judgment of the treating surgeon at any point within the study window. If this occurs, then surgeons may proceed with rescue appendectomy or percutaneous drainage in the setting of appendicitis, or with placement of a percutaneous cholecystostomy tube in the setting of acute cholecystitis.
  Arms: Non-operative management

SUMMARY:
This study evaluates operative and non-operative management of acute appendicitis (infection or inflammation of the appendix) and acute cholecystitis (inflammation/infection of the gallbladder) in patients with active mild to moderate COVID-19 infection. The hypothesis is that COVID+ patients with uncomplicated acute appendicitis or acute cholecystitis amendable to a laparoscopic procedure can have safe operative outcomes compared to those managed non-operatively.

DETAILED DESCRIPTION:
As the novel coronavirus disease 2019 (COVID-19) disseminates across the United States, more routine preoperative testing is going to expose infected patients with no or mild pneumonia symptoms. Currently, little is known regarding the true consequences of general anesthesia in COVID-positive (COVID+) patients. Surgeons are going to face challenging decisions regarding whether or not to operate for non-elective cases requiring general anesthesia when non-operative treatment options exist. Patients with acute appendicitis are usually treated with an operation to remove the appendix, but they can also be initially treated with antibiotics and have an operation at a later date. Similarly, patients with acute cholecystitis are usually treated with an operation to remove the gallbladder, but they can be treated with antibiotics and a percutaneous cholecystostomy tube (a tube that going through the skin to drain the gallbladder) and have an operation at a later date. However, patients managed without a definitive operation may require more resource utilization, PPE consumption, interactions with hospital personnel, and could experience treatment failures that exacerbate their viral illness. This is a pilot study comparing the safety of operative versus non-operative management of COVID+ patients with mild to moderate symptoms.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 confirmed positive by a microbiologic test.
* Mild COVID-19 - no or mild pneumonia
* EITHER

  1. Uncomplicated acute appendicitis without a fecalith OR
  2. Acute cholecystitis - by TG18/TG13 diagnostic criteria where definite diagnosis requires one item in A + one item in B + C A. Local signs of inflammation etc.

  <!-- -->

  1. Murphy's sign
  2. RUQ mass/pain/tenderness B. Systemic signs of inflammation etc.

  <!-- -->

  1. Fever
  2. elevated CRP
  3. elevated WBC count C. Imaging findings characteristic of acute cholecystitis

Exclusion Criteria:

* Active pregnancy
* COVID-19 severe disease that would be a contraindication to operative intervention at the discretion of the attending surgeon supported by the following, none of which are individually required or are a strict exclusion criterion as some of these could be attributed or exacerbated by the underlying surgical problem:

  1. Persistent dyspnea
  2. Persistent respiratory frequency >30/min
  3. Persistent blood oxygen saturation <93%
  4. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio <300
  5. Lung infiltrates >50%
* COVID-19 critical disease - respiratory failure, shock, or multiorgan dysfunction
* The surgeon expects increased operative complexity - high risk of conversion to open or prolonged procedure
* Unable or unwilling to consent or fulfill study procedures - need to complete 90 day follow-up by telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton C Petro, MD, Principal Investigator — Associate Professor of Surgery
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Lei S, Jiang F, Su W, Chen C, Chen J, Mei W, Zhan LY, Jia Y, Zhang L, Liu D, Xia ZY, Xia Z. Clinical characteristics and outcomes of patients undergoing surgeries during the incubation period of COVID-19 infection. EClinicalMedicine. 2020 Apr 5;21:100331. doi: 10.1016/j.eclinm.2020.100331. eCollection 2020 Apr. PMID 32292899
- [Background] Aminian A, Safari S, Razeghian-Jahromi A, Ghorbani M, Delaney CP. COVID-19 Outbreak and Surgical Practice: Unexpected Fatality in Perioperative Period. Ann Surg. 2020 Jul;272(1):e27-e29. doi: 10.1097/SLA.0000000000003925. PMID 32221117
- [Background] Podda M, Gerardi C, Cillara N, Fearnhead N, Gomes CA, Birindelli A, Mulliri A, Davies RJ, Di Saverio S. Antibiotic Treatment and Appendectomy for Uncomplicated Acute Appendicitis in Adults and Children: A Systematic Review and Meta-analysis. Ann Surg. 2019 Dec;270(6):1028-1040. doi: 10.1097/SLA.0000000000003225. PMID 30720508
- [Background] Gomi H, Solomkin JS, Schlossberg D, Okamoto K, Takada T, Strasberg SM, Ukai T, Endo I, Iwashita Y, Hibi T, Pitt HA, Matsunaga N, Takamori Y, Umezawa A, Asai K, Suzuki K, Han HS, Hwang TL, Mori Y, Yoon YS, Huang WS, Belli G, Dervenis C, Yokoe M, Kiriyama S, Itoi T, Jagannath P, Garden OJ, Miura F, de Santibanes E, Shikata S, Noguchi Y, Wada K, Honda G, Supe AN, Yoshida M, Mayumi T, Gouma DJ, Deziel DJ, Liau KH, Chen MF, Liu KH, Su CH, Chan ACW, Yoon DS, Choi IS, Jonas E, Chen XP, Fan ST, Ker CG, Gimenez ME, Kitano S, Inomata M, Mukai S, Higuchi R, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: antimicrobial therapy for acute cholangitis and cholecystitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):3-16. doi: 10.1002/jhbp.518. Epub 2018 Jan 9. PMID 29090866
- [Background] Davis CA, Landercasper J, Gundersen LH, Lambert PJ. Effective use of percutaneous cholecystostomy in high-risk surgical patients: techniques, tube management, and results. Arch Surg. 1999 Jul;134(7):727-31; discussion 731-2. doi: 10.1001/archsurg.134.7.727. PMID 10401823
- [Background] Yokoe M, Hata J, Takada T, Strasberg SM, Asbun HJ, Wakabayashi G, Kozaka K, Endo I, Deziel DJ, Miura F, Okamoto K, Hwang TL, Huang WS, Ker CG, Chen MF, Han HS, Yoon YS, Choi IS, Yoon DS, Noguchi Y, Shikata S, Ukai T, Higuchi R, Gabata T, Mori Y, Iwashita Y, Hibi T, Jagannath P, Jonas E, Liau KH, Dervenis C, Gouma DJ, Cherqui D, Belli G, Garden OJ, Gimenez ME, de Santibanes E, Suzuki K, Umezawa A, Supe AN, Pitt HA, Singh H, Chan ACW, Lau WY, Teoh AYB, Honda G, Sugioka A, Asai K, Gomi H, Itoi T, Kiriyama S, Yoshida M, Mayumi T, Matsumura N, Tokumura H, Kitano S, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: diagnostic criteria and severity grading of acute cholecystitis (with videos). J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):41-54. doi: 10.1002/jhbp.515. Epub 2018 Jan 9. PMID 29032636

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-operative Management: Treatment with antibiotics
  Non-operative management: Patients will be treated with 3 days of intravenous antibiotics followed by 7 days of oral antibiotics, as described below:
  Non-penicillin allergic patients
  * piperacillin/tazobactam 3.375g IV every 6 hours for 3 days
  * amoxicillin/clavulanate 875/125mg by mouth every 12 hours for 7 days
  Penicillin allergic patients
  * ertapenem 1g IV every 24 hours for 3 days
  * ciprofloxacin 500mg every 12 hours AND metronidazole 500mg every 8 hours for 7 days
  Patients may be considered to have failed non-operative management (e.g. treatment failure) if they experience absence of clinical improvement, worsening abdominal pain and/or localized/diffuse peritonitis in the judgment of the treating surgeon at any point within the study window. If this occurs, then surgeons may proceed with rescue appendectomy or percutaneous drainage in the setting of appendicitis, or with placement of a percutaneous cholecystostomy tube in the setting of acute cholecystitis.
Period: Overall Study
Arm/Group | Operative Management | Non-operative Management
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Operative Management | Non-operative Management | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Median (Full Range); unit: Years] | 32 [32 to 32] | 72 [72 to 72] | 52 [32 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pulmonary Complications
Description: Including pneumonia, acute respiratory distress syndrome (ARDS) or unexpected postoperative ventilation
  For operative management this means any episode of non-invasive ventilation, invasive ventilation, or extracorporeal membrane oxygenation after initial extubation after surgery, or patient cannot be extubated as planned after surgery.
  For non-operative management this means any intubation
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Operative Management | Non-operative Management
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With Post-intervention ICU Admission
Description: ICU admission following randomization
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Operative Management | Non-operative Management
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

3. Secondary Outcome: Mortality (All Cause)
Description: Any death
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Operative Management | Non-operative Management
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

4. Secondary Outcome: Complications as Measured by the Clavien-Dindo Classification
Description: The Clavien-Dindo classification is a grading scale from 1 to 5 (with 5 being more severe0 to objectively describe the severity of a complication, including any deviation from the normal postoperative course
Time Frame: Up to 90 days
Population: Subject in the Operative management did not develop any complications that met Clavien-Dindo classification
Measure: Number; unit: score on a scale
Arm/Group | Non-operative Management
Number analyzed (Participants) | 1
score on a scale | 1

5. Secondary Outcome: Median Length of Hospital Stay
Description: Cumulative and individual length of hospitalization(s)
Time Frame: Up to 90 days
Measure: Number; unit: Hours
Arm/Group | Operative Management | Non-operative Management
Number analyzed (Participants) | 1 | 1
Hours | 44 | 137

6. Secondary Outcome: Number of Emergency Room Visits/Readmission
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Operative Management | Non-operative Management
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Treatment Failure for Non-operative Management
Description: Patients randomized to non-operative management who require non-elective surgery to remove the affected organ
Time Frame: Up to 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Operative Management
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: 90 days following intervention
Arm/Group | Operative Management | Non-operative Management
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT04748120/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT04748120/ICF_001.pdf